CLINICAL TRIAL: NCT07368218
Title: Randomized Clinical Trial on Morbidity, Psychological Impact, and Changes in Biomarker Concentration During the Perioperative Period Comparing Transmesocolic Versus Retromesenteric Reconstruction in Cephalic Duodenopancreatectomy (FAST Trial)
Brief Title: Comparison of Transmesocolic Versus Retromesenteric Reconstruction in Cephalic Duodenopancreatectomy (FAST Trial)
Acronym: FAST
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Universitari de Bellvitge (Other)
Responsible Party: Principal Investigator, BUSQUETS, JULI, Head of Pancreatic Surgery Unit, Hospital Universitari de Bellvitge
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: HUB-CIR-FAST
Record Dates: First submitted 2026-01-11; First posted 2026-01-26 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Pancreatic Cancer
Keywords: duodenopancreatectomy; Pancreatic cancer; Delayed Gastric emptying
MeSH Terms: conditions — Pancreatic Neoplasms; Gastroparesis

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Retromesenteric reconstruction (Experimental)
  Interventions: Procedure: Retromesenteric reconstruction
- Transmesocolic reconstruction (Active Comparator)
  Interventions: Procedure: Transmesocolic reconstruction

INTERVENTIONS:
Procedure: Retromesenteric reconstruction — Perform a retromesenteric reconstruction after pancreaticoduodenectomy
  Arms: Retromesenteric reconstruction
Procedure: Transmesocolic reconstruction — Perform the standard reconstruction procedure (transmesocolic) pancreaticoduodenectomy
  Arms: Transmesocolic reconstruction

SUMMARY:
Objective: To compare the incidence of delayed gastric emptying (ISGPS 2007 criteria) between patients undergoing retromesenteric versus transmesocolic reconstruction after pancreaticoduodenectomy. Secondary objectives include evaluating overall postoperative morbidity (Clavien-Dindo ≥ Grade I) at 90 days, postoperative pancreatic fistula according to ISGPF criteria, 30- and 90-day mortality, differences in operative time and blood loss, hospital stay duration, exploratory analysis of inflammatory biomarkers in serum and drainage fluid, psychological impact using SCL-90-R scale, and postoperative quality of life using EORTC QLQ-C30 scale.

Methods: Randomized, controlled, single-center superiority clinical trial with 1:1 allocation. One hundred twenty-four patients candidates for duodenopancreatectomy due to pancreatic pathology will be randomized using balanced blocks to transmesocolic (control) or retromesenteric (study) reconstruction. Randomization will be revealed after completing the resection phase. Primary intention-to-treat analysis will estimate relative risk with 95% CI for dichotomous variables, Kaplan-Meier survival analysis with log-rank test, and linear mixed models for repeated measures in quality of life outcomes. Follow-up will be 90 days for the primary endpoint, extending to 12 months for secondary objectives.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Candidates for cephalic duodenopancreatectomy due to pancreatic pathology
* Ability to complete follow-up questionnaires

Exclusion Criteria:

* Emergency surgery
* Participation in another clinical trial
* Pregnancy or lactation
* Severe psychiatric disorder that prevents follow-up
* Inability to understand the information and sign study consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 124 (Estimated)
Dates: Start 2026-01-31 (Estimated); Primary Completion 2027-06 (Estimated); Study Completion 2028-06 (Estimated)

PRIMARY OUTCOMES:
Delayed Gastric Emptying | From first postoperative day to 30 days
  Delayed gastric emptying according to ISGPS 2007 definition: Grade A (nasogastric tube >3 days or reinsertion between days 4-7 + vomiting); Grade B (tube >7 days or reinsertion after day 7 + vomiting); Grade C (impossibility of oral tolerance after day 14)

SECONDARY OUTCOMES:
Postoperative morbility | Form first postoperative day to day 30
  Postoperative morbidity at 90 days according to Clavien-Dindo classification (≥ Grade I)
Pancreatic fistula | From first postoperative day to day 30
  Pancreatic fistula according to ISGPF 2016 definition: Grade A (drainage amylase >3x normal on day 3 without clinical impact); Grade B (requiring management change); Grade C (reintervention or death)
Mortality | From first postoperative day to day 90
  30- and 90-day mortality (any cause)
Hospital stay | From first postoperative day to hospital discharge up to 15 weeks
  Postoperative hospital stay days (from surgery to hospital discharge)
Operative time | Periprocedural time, an average time of 300-400 minutes
  Total operative time (minutes)
Proportion of patients with NLR index ≥5 | From the first postoperative day to one year follow-up
  First, a preoperative NLR index determination from the preoperative blood count.
  Proportion of patients with NLR cut-off point ≥5, which is associated with lower overall survival and recurrence-free survival in patients undergoing pancreatic resection.
Proportion of patients with CA19.9 >37 U/ml | From the first postoperative day to one year follow-up
  First, a preoperative CA19.9 measurement from preoperative laboratory tests. Determination of the proportion of patients with CA 19.9 cut-off point >37 U/ml, as it is considered elevated according to the standard reference range.
Cytokines in serum | From the first postoperative day to day 90
  * Cytokine concentration in serum: continuous variable measured at 24 hours and day 5 post-surgery in a subsample of 30 patients.
  * Detection panel: 2000 inflammatory biomarkers using high-sensitivity semi-quantitative Raybiotech L-series arrays with densitometric reading
Cytokines in abdominal drainage | From the first postoperative day to day 90
  * Cytokine concentration in drainage fluid: continuous variable measured at 24 hours and day 5 post-surgery in a subsample of 30 patients.
  * Detection panel: 2000 inflammatory biomarkers using high-sensitivity semi-quantitative Raybiotech L-series arrays with densitometric reading
Cytokines and complications correlation | From the first postoperative day to day 90
  Exploratory analysis of the association between cytokine levels and the appearance of complications during the first 90 days.
Recurrence | From the first postoperative day to one year follow-up
  - Recurrence of malignant pathology: Defined as the appearance of local, regional, or distant disease documented by imaging techniques (CT/MRI) or histopathological confirmation.
Time to recurrence | From the first postoperative day to one year follow-up
  - Time to recurrence: Time elapsed from surgery to detection of recurrence (months).
Complications-recurrence correlation | From the first postoperative day to one year follow-up
  Association analysis between the presence of complications (Clavien-Dindo ≥ II) and early recurrence (≤12 months).

CONTACTS AND LOCATIONS:
Locations (1):
- Hopital Universitari de Bellvitge, L'Hospitalet de Llobregat, Spain, Spain

IPD SHARING:
Plan to Share IPD: No